CLINICAL TRIAL: NCT01972854
Title: A Multi-Center, Randomized, Placebo-Controlled Evaluation of the Safety and Efficacy of the KXL System With VibeX (Riboflavin Ophthalmic Solution) for Corneal Collagen Cross-Linking in Eyes With Keratoconus
Brief Title: Safety and Efficacy of Corneal Collagen Cross-Linking in Eyes With Keratoconus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KXL-005
Record Dates: First submitted 2013-10-25; First posted 2013-10-31 (Estimated); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Keratoconus
Keywords: keratoconus; cross-linking; KXL
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- riboflavin solution and KXL System (Experimental): The cornea will receive 5 drops of VibeX (0.12% riboflavin ophthalmic solution). Five additional VibeX drops will be instilled every two minutes for 20 minutes. The eye will be irradiated for 8 minutes with an on/off cycle of 1 second UVA on/1 second UVA off.
  Interventions: Drug: riboflavin solution; Device: KXL System
- placebo solution and KXL System (Placebo Comparator): The cornea will receive 5 drops of placebo (0.0% riboflavin ophthalmic solution. Five additional placebo drops will be instilled every two minutes for 20 minutes. The eye will be irradiated for 8 minutes with an on/off cycle of 1 second UVA on/1 second UVA off.
  Interventions: Drug: placebo solution; Device: KXL System

INTERVENTIONS:
Drug: riboflavin solution — 0.12% riboflavin ophthalmic solution
  Other Names: VibeX
  Arms: riboflavin solution and KXL System
Drug: placebo solution — 0.0% riboflavin ophthalmic solution
  Other Names: placebo
  Arms: placebo solution and KXL System
Device: KXL System — 30mW/cm2
  Other Names: UVA Irradiation

SUMMARY:
The objectives of this study are to evaluate the safety and efficacy of corneal collagen cross-linking performed with VibeX (riboflavin ophthalmic solution) and the KXL System as compared to placebo in impeding the progression of, and/or reducing, maximum corneal curvature.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria in order to be enrolled in the trial:

1. Be at least 12 years of age, male or female, of any race;
2. Provide written informed consent and sign a HIPAA form. Subjects who are under the age of 18 (or have not yet reached the age of majority per local regulations) will need to sign an assent form as well as having a parent or legal guardian sign an informed consent;
3. Willingness and ability to follow all instructions and comply with schedule for follow-up visits, including the ability to read English to complete the NEI-VFQ 25 questionnaire;
4. For females capable of becoming pregnant, agree to have urine pregnancy testing performed at Visit 2 prior to randomization of the study eye and prior to treatment of a fellow and/or cross-over eye; must not be lactating, and must agree to use a medically acceptable form of birth control for at least one week prior to Visit 2, one week prior to treatment of a fellow eye or cross-over eye, and continue to use the method for one month following the last treatment. Acceptable forms for birth control are spermicide with barrier, oral contraceptive, injectable or implantable method of contraception, transdermal contraceptive, intrauterine device, or surgical sterilization of partner. For non-sexually active females, abstinence will be considered an acceptable form of birth control. Women considered capable of becoming pregnant include all females who have experienced menarche and have not experienced menopause (as defined by amenorrhea for greater than 12 consecutive months) or have not undergone successful surgical sterilization (e.g. hysterectomy, bilateral tubal ligation, or bilateral oophorectomy);
5. Subjects > 25 years old at the time of screening of their study eye must meet the following criteria. Subjects ≤ 25 years old and all subjects who have their fellow-eye or crossover eye treated are not required to meet these criteria;

   - Having a diagnosis of progressive keratoconus defined as one or more of the following changes over a period of 36 months or less:
   1. An increase of ≥ 1.00 D in the steepest keratometry value (ksteep)
   2. An increase of ≥ 1.00 D in regular astigmatism evaluated by subjective manifest refraction or as evaluated by comparing eyeglass or contact lens prescriptions to current subjective manifest refraction
   3. A myopic shift (decrease in the spherical equivalent) of ≥ 0.50 D in subjective manifest refraction or as evaluated by comparing eyeglass or contact lens prescriptions to current subjective manifest refraction
   4. A decrease ≥ 0.1 mm in the BOZR (Back Optical Zone Radius) in rigid contact lens wearers where other information is not available
6. Having topographic evidence of keratoconus with a diagnosis of mild, moderate, or severe keratoconus defined as the following:

   * Mild Keratoconus:

     1. Axial topography consistent with keratoconus
     2. Flat Pentacam keratometry reading ≤ 51.00D
   * Moderate Keratoconus:

     1. Axial topography consistent with keratoconus
     2. Flat Pentacam keratometry reading > 51.00 D and ≤ 56.00 D or astigmatism ≥ 8.00 D
   * Severe Keratoconus:

     1. Axial topography consistent with keratoconus with marked areas of steepening
     2. Flat Pentacam keratometry reading > 56.00 D
7. Presence of central or inferior steepening on the Pentacam map;
8. Have a maximum corneal curvature, as measured by Kmax, of ≥ 47.00 D;
9. BSCVA of ≥ 1 letter and ≤ 80 letters on ETDRS chart;
10. Contact Lens Wearers Only: Removal of contact lenses is required for a 1 week period prior to the first screening refraction visit (and each subsequent Visit 1, as necessary) and must remain out until the 1 month visit is completed;
11. Contact Lens Wearers Only: Manifest refraction must be stable between two consecutive visits which occur at least 7 days apart. A stable refraction is one in which the manifest refraction spherical equivalent and the average K (Km) on the Pentacam taken at the first visit do not differ by more than 0.75 D from the respective measurements taken at the second exam. A contact lens wearer is defined as someone who has worn contact lenses in the eye to be treated in the last 30 days.

Exclusion Criteria:

Subjects must not meet any of the following criteria to be enrolled in the trial:

1. Contraindications, sensitivity or known allergy to the use of the test article(s) or their components;
2. If female, be pregnant, nursing or planning a pregnancy during the course of the study or have a positive urine pregnancy test at Visit 2 prior to randomization or treatment of either eye;
3. Eyes classified as either normal, atypical normal, or keratoconus suspect on the severity grading scheme;
4. A history of previous corneal surgery or the insertion of Intacs in the eye to be treated;
5. A history of previous Limbal Relaxing Incision (LRI) procedure in the eye to be treated;
6. Corneal pachymetry that is < 375 microns prior to epithelial debridement at the thinnest point measured by Pentacam in the eye to be treated;
7. Eyes which are aphakic;
8. Eyes which are pseudophakic and do not have a UV blocking lens implanted;
9. Previous ocular condition (other than refractive error) in the eye to be treated that may predispose the eye for future complications. For example:

   1. History or evidence of active or inactive corneal disease (e.g., herpes simplex keratitis, herpes zoster keratitis, corneal melt, recurrent corneal erosion syndrome, corneal dystrophy, etc.);
   2. Clinically significant corneal scarring in the cross-linking treatment zone that is not related to keratoconus or, in the investigator's opinion, will interfere with the cross-linking procedure;
10. A history of delayed epithelial healing in the eye to be treated;
11. Subjects with nystagmus or any other condition that would prevent a steady gaze during the treatment or other diagnostic tests;
12. Subjects with a current condition that, in the investigator's opinion, would interfere with or prolong epithelial healing;
13. Taking supplements containing Vitamin C (ascorbic acid) within 1 week of the cross-linking treatment;
14. A history of previous corneal crosslinking treatment in the eye to be treated;
15. The subject should not have participated in any investigational drug or device study within 30 days of screening or be concurrently enrolled in another investigational drug or device study.
16. The Investigator may exclude or discontinue any subject for any sound medical reason.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2013-11; Primary Completion 2016-03 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in Kmax from baseline | 12 months
  The primary endpoint is the mean change from baseline to 12 months in maximum corneal curvature (Kmax) between the VibeX treatment group and the Placebo control group.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hersh, M.D., Study Director — Glaukos Corporation
Locations (11):
- United States (11):
  - UC Irvine Department of Ophthalmology, Irvine, California
  - Gordon -Weiss Vision Institute, San Diego, California
  - Price Vision Group, Indianapolis, Indiana
  - Durrie Vision, Overland Park, Kansas
  - Ophthalmic Consultants of Boston, Waltham, Massachusetts
  - Hersh Vision Group, Teaneck, New Jersey
  - UPMC Eye Center, Pittsburgh, Pennsylvania
  - Vance Thompson Vision, Sioux Falls, South Dakota
  - Focal Point Vision, San Antonio, Texas
  - Hoopes Vision, Draper, Utah
  - See Clearly Vision, McLean, Virginia

IPD SHARING:
Plan to Share IPD: No